CLINICAL TRIAL: NCT01655017
Title: Fibrosis a New Pathological Actor in Adipose Tissue
Acronym: fibrota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P100503
Record Dates: First submitted 2012-04-25; First posted 2012-08-01 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Metabolic Diseases; Fibrosis; Body Weight
Keywords: Obesity; adipose tissue fibrosis; Adipose tissue inflammation; Low grade systemic inflammation; non invasive device; Bariatric surgery
MeSH Terms: conditions — Obesity; Metabolic Diseases; Fibrosis; Body Weight | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- biopsy (Experimental): Obesity with BMI> 40 kg/m² or obesity with BMI between >35 kg/m² with comorbidities (OSA, type 2 diabetes, hypertension etc…)
  Interventions: Procedure: biopsy
- healthy volunteers (No Intervention): biopsy during a surgery

INTERVENTIONS:
Procedure: biopsy — adipose tissue biopsy (to evaluate inflammation and fibrosis)
  Arms: biopsy

SUMMARY:
Adipose tissue (AT) has specific alterations in obesity in particular increased fibrosis amount compared to lean subjects. Fibrosis amount measured by immunohistochemistry on adipose biopsies appears to to predict weight loss response after a bariatric surgery. Non invasive tools to measure fibrosis needs to be validated. The investigators primary aim is to validate a new device able to measure adipose tissue stiffness.

Thus the investigators plan to compare the stiffness results obtained with the device to the quantification of fibrosis using immuno-chemistry in massively obese patient's candidates to a bariatric surgery.

DETAILED DESCRIPTION:
Adipose tissue (AT) has specific alterations in obesity that could link obesity to its comorbidities. In particular increased fibrosis abundance in AT has been observed in obese compared to lean subjects. The investigators previously observed that the amount of fibrosis in AT measured at baseline could predict surgery-induced weight loss. Patient with the higher amount of fibrosis at baseline were those who lost less fat mass one year after surgery.

To date fibrosis can only be measured using by immunohistochemistry after surgical biopsy. To that prospect, non invasive tools need to be validated, in particular device able to measure adipose tissue stiffness. The investigators hypothesis is that this new device is as powerful as IHC-quantified fibrosis to predict surgery induced weight loss.

To answer that question the investigators will evaluate adipose tissue stiffness with the device as well as quantify fibrosis using immuno-chemistry on AT biopsy in morbidly obese patients before and during the first year after a bariatric surgery.

The first objective is to validate the investigators new device by comparing both invasive fibrosis measurement on adipose tissue and non invasive stiffness measure The investigators second objective is to assess whether the investigators device can predict weight loss repose after bariatric surgery.

This project is based on a clinical protocol performed in massively obese subjects (BMI>40 kg/m² or BMI>35kg/m² with comorbidities). The investigators will recruit 250 obese patients addressed for bariatric surgery (bypass, sleeve or gastric banding). Clinical phenotype, biochemical analysis, body composition, systemic inflammation, adipose tissue biopsy (to evaluate inflammation and fibrosis) will be assessed at baseline and 3 and 12 months after surgery. Also at baseline surgical sub cutaneous and omental adipose tissue (to evaluate inflammation and fibrosis) as well as liver biopsy (to score non alcoholic hepatitis) will be analysed. 50 non obese patients will serve as controls. Adipose tissue stiffness measured with the device as well as fibrosis quantification on subcutaneous and omental adipose tissue will be assessed at baseline during programmed non inflammatory abdominal surgery Associations between all clinical and biological parameters will be assessed at the different point of the follow up.

More generally, this project might lead us to elucidate whether fibrosis in adipose tissue can predict surgery outcome in terms of weight loss and obesity related complications improvement. Also the investigators want to validate a new non invasive tool to measure adipose tissue fibrosis and check whether it can predict surgery outcomes.

ELIGIBILITY:
Inclusion criteria :

Obese population :

* Obesity with BMI> 40 kg/m² or obesity with BMI >35 kg/m² with comorbidities (OSA, type 2 diabetes, hypertension etc…)
* Age: 18-65
* weight stable for three months preceding surgery
* candidate to a sleeve or bypass or adjustable gastric banding

Controls:

* BMI< 30 kg/m²
* Age: 18-65
* non inflammatory acute or chronic disease
* candidate to a programmed non inflammatory abdominal surgery

Exclusion criteria :

* Inflammatory disease
* Pregnancy
* cancer
* Drugs (AINS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2012-02-08 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Adipose tissue stiffness and fibrosis | baseline
  In both massively obese patients and in a subgroup of lean and overweight control, adipose tissue stiffness will be assessed using the elastography non invasive device. Adipose tissue fibrosis will be evaluated using immuno-chemistry staining upon adipose tissue surgical biopsy and defined as the ratio of the surface stained with picrosirius and the surface of the biopsy. The investigators will then look for a strong statistical association between those two measures to validate our new device.

SECONDARY OUTCOMES:
weight loss one year after surgery | 12 months
  The investigators will separate our massively obese patients in tertiles upon weight loss importance one year after surgery and evaluate whether those who lose the most important amount of weight are those who had the less adipose tissue stiffness before the surgery
Severity of obesity related disease before surgery (in particular NASH acknowledged on liver histology) | baseline
  The investigators will evaluate whether we find a significant correlation between the severity of obesity related disease and the adipose tissue stiffness at baseline.
Obesity related disease improvement one year after surgery. | 12 months
  The investigators will check whether patients with the less important adipose tissue stiffness are those who improve the most their obesity related disease (separating our population in two those who improve and those who don't)
Adipose tissue fibrosis and weight loss response | 3 months
  The investigators will quantify adipose tissue fibrosis using picrosirius staining on surgical adipose tissue and evaluate whether the amount of fibrosis at three months negatively correlates with weight loss.
Adipose tissue stiffness and weight loss response | 3 months
  The investigators will quantify adipose stiffness using the non invasive device and evaluate whether the severity of adipose stiffness at three months negatively correlates with weight loss.
Adipose tissue fibrosis and weight loss response. | 12 months
  The investigators will quantify adipose tissue fibrosis using picrosirius staining on surgical adipose tissue and evaluate whether the amount of fibrosis at 12 months negatively correlates with weight loss.
Adipose tissue stiffness and the severity of obesity related disease. | 3 months
  evaluate whether the patients who improve the most their obesity related disease in the short term are those who decreases the most their adipose stiffness.
Adipose tissue stiffness and the severity of obesity related disease. | 12 months
  evaluate whether the patients who improve the most their obesity related disease in the long term are those who decreases the most their adipose stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aron-wisnewsky, MD, Principal Investigator — APHP; Karine Clement, MD, PhD, Study Director — APHP
Locations (2):
- France (2):
  - Service de Chirurgie générale et digestive et d'oncologie du Pr Nordlinger -Ambroise Paré, Boulogne
  - Service de nutrition du Pr Basdevant -Pitié salpêtrière/ Institut Cardiometabolism and nutrition, Paris

REFERENCES:
- [Derived] Torres L, Camila Goncalves Miranda M, Dantas Martins V, Caixeta F, de Almeida Oliveira M, Martins Trindade L, Carvalho de Assis H, Nascimento V, Pinheiro Rosa N, Gomes E, Oliveira Almeida S, Marquet F, Genser L, Marcelin G, Clement K, Russo M, Maria Caetano Faria A, Uceli Maioli T. Obesity-induced hyperglycemia impairs oral tolerance induction and aggravates food allergy. Mucosal Immunol. 2023 Aug;16(4):513-526. doi: 10.1016/j.mucimm.2023.05.008. Epub 2023 Jun 10. PMID 37302712
- [Derived] Bel Lassen P, Nori N, Bedossa P, Genser L, Aron-Wisnewsky J, Poitou C, Surabattula R, Juul Nielsen M, Asser Karsdal M, Julie Leeming D, Schuppan D, Clement K. Fibrogenesis Marker PRO-C3 Is Higher in Advanced Liver Fibrosis and Improves in Patients Undergoing Bariatric Surgery. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1356-e1366. doi: 10.1210/clinem/dgab897. PMID 34905051
- [Derived] Rouault C, Marcelin G, Adriouch S, Rose C, Genser L, Ambrosini M, Bichet JC, Zhang Y, Marquet F, Aron-Wisnewsky J, Poitou C, Andre S, Derumeaux G, Guerre-Millo M, Clement K. Senescence-associated beta-galactosidase in subcutaneous adipose tissue associates with altered glycaemic status and truncal fat in severe obesity. Diabetologia. 2021 Jan;64(1):240-254. doi: 10.1007/s00125-020-05307-0. Epub 2020 Oct 30. PMID 33125520
- [Derived] Bel Lassen P, Charlotte F, Liu Y, Bedossa P, Le Naour G, Tordjman J, Poitou C, Bouillot JL, Genser L, Zucker JD, Sokolovska N, Aron-Wisnewsky J, Clement K. The FAT Score, a Fibrosis Score of Adipose Tissue: Predicting Weight-Loss Outcome After Gastric Bypass. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2443-2453. doi: 10.1210/jc.2017-00138. PMID 28419237
- [Derived] Liu Y, Aron-Wisnewsky J, Marcelin G, Genser L, Le Naour G, Torcivia A, Bauvois B, Bouchet S, Pelloux V, Sasso M, Miette V, Tordjman J, Clement K. Accumulation and Changes in Composition of Collagens in Subcutaneous Adipose Tissue After Bariatric Surgery. J Clin Endocrinol Metab. 2016 Jan;101(1):293-304. doi: 10.1210/jc.2015-3348. Epub 2015 Nov 19. PMID 26583585
- [Derived] Verger EO, Aron-Wisnewsky J, Dao MC, Kayser BD, Oppert JM, Bouillot JL, Torcivia A, Clement K. Micronutrient and Protein Deficiencies After Gastric Bypass and Sleeve Gastrectomy: a 1-year Follow-up. Obes Surg. 2016 Apr;26(4):785-96. doi: 10.1007/s11695-015-1803-7. PMID 26205215